CLINICAL TRIAL: NCT05058053
Title: INVESTIGATION OF THE EFFECT OF COLD APPLICATION ON THE DEVELOPMENT OF PHLEBITIS IN PATIENTS RECEIVING INTRAVENOUS AMIODARONE TREATMENT. A RANDOMIZED OPEN-LABEL TRIAL
Brief Title: THE EFFECT OF COLD APPLICATION ON THE DEVELOPMENT OF PHLEBITIS IN PATIENTS RECEIVING INTRAVENOUS AMIODARONE TREATMENT.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Tulay Basak, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 788
Record Dates: First submitted 2021-09-07; First posted 2021-09-27 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Phlebitis
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold application group (Experimental): After starting amiodarone treatment, cold application was applied a total of 12 times on the infused PVC with cold gel packs for 15 minutes at 2-hour intervals. At all stages of the study, the researcher closely monitored the patients. During the treatment, the development of phlebitis after cold application during the 24-hour infusion was evaluated every 2 hours by the researcher using the "Visual Infusion Phlebitis Scale" and recorded. After starting the amiodarone infusion, the patients were observed for the development of phlebitis for 24 hours until the end of the procedure and for 2 hours after the end of the treatment.
  Interventions: Other: Cold application
- Control group (No Intervention): the patients who were started on amiodarone infusion were observed for the development of phlebitis, receiving no intervention. During the treatment, phlebitis development was evaluated and recorded by the researcher using the "Visual Infusion Phlebitis Scale" every 2 hours during the 24-hour infusion. After starting the amiodarone infusion, the patients were observed for the development of phlebitis for 24 hours until the end of the procedure and for 2 hours after the end of the treatment.

INTERVENTIONS:
Other: Cold application — Cold application was applied a total of 12 times on the infused PVC with cold gel packs for 15 minutes at 2-hour intervals.
  Arms: Cold application group

SUMMARY:
This study, which has a quasi-experimental, prospective, and open-label randomized controlled design, was conducted to examine the effect of cold application on the development of phlebitis in patients receiving IV amiodarone infusion treatment.

Study Hypotheses H0-1: There is no difference in the rate of development of phlebitis between the patients who received and who did not receive cold application during amiodarone IV infusion.

H0-2: There is no difference in the grade of phlebitis between the patients who received and who did not receive cold application during amiodarone IV infusion.

H0-3: There is no difference in the time of development of phlebitis between the patients who received and who did not receive cold application during amiodarone IV infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18, who were planned to receive 300 mg amiodarone in 150 ccs of 5% dextrose + 900 mg amiodarone (maintenance) in 50 ccs of 5% Dextrose in 30 minutes (24 hour-infusion),
* Patients to whom PVC was placed in the upper extremity, and who did not develop phlebitis on the PVC site

Exclusion Criteria:

* Cold allergy/sensitivity or circulatory disorders
* During the study, patients who had a change in the IV amiodarone treatment protocol, whose IV amiodarone treatment was terminated before 24 hours, whose IV amiodarone treatment protocol was started, but PVC had to be replaced for any reason during the 24-hour period

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
the rate of development of phlebitis | 24+2 hours
  the patients were observed for the development of phlebitis for 24 hours until the end of the procedure and for 2 hours after the end of the treatment.During the treatment, the development of phlebitis after cold application during the 24-hour infusion was evaluated every 2 hours by the researcher using the "Visual Infusion Phlebitis Scale" and recorded.

SECONDARY OUTCOMES:
the grade of phlebitis | 24+2 hours
  the patients were observed for the development of phlebitis for 24 hours until the end of the procedure and for 2 hours after the end of the treatment.During the treatment, the development of phlebitis after cold application during the 24-hour infusion was evaluated every 2 hours by the researcher using the "Visual Infusion Phlebitis Scale" and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okyay B, Basak T. The effect of cold gel pack application in the prevention of amiodarone-related phlebitis. Nurs Crit Care. 2024 Nov;29(6):1739-1743. doi: 10.1111/nicc.13020. Epub 2024 Jan 30. PMID 38290741